CLINICAL TRIAL: NCT02922998
Title: Monitoring CD64 on Neutrophils Regarding Effects of Antibiotics in Patients With SIRS Developing Sepsis
Brief Title: CD64 and Antibiotics in Human Sepsis
Acronym: CD64SEPLDX
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, University of Ulm
Other Study IDs: LeukoDx_CD64_AB_sepsis
Record Dates: First submitted 2016-09-26; First posted 2016-10-04 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Antibiotic Resistant Infection; Critical Illness; SIRS; Sepsis
Keywords: CD64 antigens; Biomarkers; Granulocyte Colony-Stimulating Factor; Interleukin-4; Interferon-gamma; C-reactive protein; lipopolysaccharide-binding protein; procalcitonin; Cytokines; Patients; Human; Systemic Inflammatory Response Syndrome; Sepsis; Infection; Antibiotics; Intensive Care Units; Point-of-Care Systems; Bedside Testing
MeSH Terms: conditions — Critical Illness; Sepsis; Systemic Inflammatory Response Syndrome; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to find out whether CD64 expression on neutrophils measured by a new bedside test (LeukoDx) within 30 minutes is associated with effective antibiotic therapy in critically ill adult patients at risk of sepsis.

DETAILED DESCRIPTION:
In the present study, in critically ill patients with suspected infection undergoing application of antibiotics, CD64 and inflammatory plasma markers will be determined on days 1 to 4.

CD64 expression on the surface of neutrophils will be determined by fluorescence activated cell sorter (FACS) and with a new bedside test (LeukoDx).

The purpose of the study is to clarify:

1. Is CD64 expression on neutrophils associated with effective antibiotic therapy in critically ill adult patients at risk of sepsis?
2. Is CD64 expression associated with distinct plasma parameters of inflammation?
3. Do the results of the gold standard CD64 determination by FACS correlate with those of a new bedside test (LeukoDx)?

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* critically ill adult patients
* sepsis
* SIRS
* initiation of antibiotic treatment
* patients < 48 hours after admission on ICU

Exclusion Criteria:

* multiple admissions on ICU, (>1 in last 2 weeks period)
* leukopenia < 1 G/l
* and thrombocytopenia
* rhG-CSF or IFN-gamma therapy up to 1 week before inclusion
* participation in another study receiving drugs or biological within the preceeding 30 days
* recent longterm corticosteroid treatment
* HIV
* patients after organ transplantation treated with immunomodulating drugs
* pregnant patients or after delivery
* life expectancy < 24 hours
* polytraumatized patients with reanimation on scene, or infest prognosis
* patients under high dose corticosteroids or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients with SIRS at risk of sepsis with suspected infections in whom application of antibiotics is started
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
CD64 expression on neutrophils measured by LeukoDx | 1 year

SECONDARY OUTCOMES:
Association of course of CD64 expression with effective antibiotic treatment | 1 year

OTHER OUTCOMES:
CD64 expression on neutrophils measured by FACS | 1 year
Association of CD64 expression with inflammatory markers | 1 year
Association of CD64 expression with cell surface markers on monocytes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, Principal Investigator — Department of Anaesthesiology, University Hospital Ulm; Ulm, Germany 89075
Locations (1):
- Department of Anaesthesiology, University Hospital Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barth E, Fischer G, Schneider EM, Wollmeyer J, Georgieff M, Weiss M. Differences in the expression of CD64 and mCD14 on polymorphonuclear cells and on monocytes in patients with septic shock. Cytokine. 2001 Jun 7;14(5):299-302. doi: 10.1006/cyto.2001.0880. PMID 11444911
- [Background] Barth E, Fischer G, Schneider EM, Moldawer LL, Georgieff M, Weiss M. Peaks of endogenous G-CSF serum concentrations are followed by an increase in respiratory burst activity of granulocytes in patients with septic shock. Cytokine. 2002 Mar 7;17(5):275-84. doi: 10.1006/cyto.2002.1010. PMID 12027409
- [Background] Weiss M, Gross-Weege W, Schneider M, Neidhardt H, Liebert S, Mirow N, Wernet P. Enhancement of neutrophil function by in vivo filgrastim treatment for prophylaxis of sepsis in surgical intensive care patients. J Crit Care. 1995 Mar;10(1):21-6. doi: 10.1016/0883-9441(95)90027-6. PMID 7538851
- [Background] Weiss M, Gross-Weege W, Harms B, Schneider EM. Filgrastim (RHG-CSF) related modulation of the inflammatory response in patients at risk of sepsis or with sepsis. Cytokine. 1996 Mar;8(3):260-5. doi: 10.1006/cyto.1996.0035. PMID 8833041
- [Background] Fischer G, Schneider EM, L Moldawer LL, Karcher C, Barth E, Suger-Wiedeck H, Georgieff M, Weiss M. CD64 surface expression on neutrophils is transiently upregulated in patients with septic shock. Intensive Care Med. 2001 Dec;27(12):1848-52. doi: 10.1007/s00134-001-1135-z. Epub 2001 Nov 8. PMID 11797018